CLINICAL TRIAL: NCT00270127
Title: Double-Blind, Placebo-Controlled Study to Assess the Effect of Early Intervention and/or Treatment With Epoetin Alfa on Anemia in Cancer Patients Receiving Non-Platinum-Containing Chemotherapy
Brief Title: Epoetin Alfa for Anemia in Patients With Cancer Receiving Non-platinum Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005917
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-01

CONDITIONS: Anemia; Cancer; Neoplasm
Keywords: Anemia; cancer; quality of life; chemotherapy; hemoglobin; transfusion; epoetin alfa; epoetin; erythropoietin
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the effectiveness of epoetin alfa versus placebo in reducing or preventing the need for transfusions in anemic patients with non-myeloid cancer on non-platinum chemotherapy, and to investigate quality-of-life benefits associated with the use of epoetin alfa. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
Cancer patients often experience anemia due to the disease itself, chemotherapy, or both. Quality of life is also affected, due in part to the fatigue associated with anemia. Previous studies with epoetin alfa have suggested that achieving a higher hemoglobin level may improve quality of life and help patients live longer. This is a randomized, double-blind, placebo-controlled, multicenter study to assess the effect of treatment with epoetin alfa in reducing or preventing anemia and transfusions in patients receiving non-platinum chemotherapy for non-myeloid cancers. The study also aims to determine whether changes in erythropoietin and hemoglobin levels after 2 weeks, serum ferritin (iron) levels after 2 weeks and changes in hemoglobin and developing red blood cells after either 2 or 4 weeks predict responsiveness to epoetin alfa. There will be 2 treatment groups: one group will receive subcutaneous epoetin alfa injections 3 times per week (starting at 150 units per kilogram, adjusted if needed to a maximum of 300 units per kilogram) and the other group will receive an equal volume of matching subcutaneous placebo. Treatment is to continue for 12 to 24 weeks (3 to 6 chemotherapy cycles), plus 4 weeks post-chemotherapy. Patients in the study will be observed a year after the study ends for survival data. The primary measure of effectiveness will be determined by the number of patients who are transfused, depending on primary tumor type (solid or blood) and level of hemoglobin (above or below 10.5 grams per deciliter). Additional measures of effectiveness include the change in hemoglobin, hematocrit, and developing red blood cells from the start of the study until study completion, and the change in quality of life. Safety evaluations (incidence and severity of adverse events, laboratory tests, vital signs and physical examinations) will be performed throughout the study. The hypothesis of the study is that epoetin alfa will be superior to placebo in reducing the need for transfusions and in improving anemia and quality of life. 150 units per kilogram of epoetin alfa (or placebo) 3 times weekly subcutaneously for 4 weeks, then continuing this dose or 300 units per kilogram, depending on developing red blood cell counts and/or hemoglobin. Study duration is 12 to 24 weeks (3 to 6 cycles) plus 4 weeks post-chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of non-myeloid malignancy
* undergoing treatment with non-platinum-containing chemotherapy, or non-platinum-containing chemotherapy is imminent
* Eastern Cooperative Oncology Group (which is a scale used by researchers to represent the level of activity that a patient is capable of) score of 0 (fully active, no disease restriction) to 3 (capable of only limited self-care, confined to bed or chair more than 50% of waking hours)
* life expectancy of at least 6 months
* baseline hemoglobin <= 10.5 grams per deciliter (or a fall in hemoglobin level >= 1.5 grams per deciliter per cycle or per month since the beginning of the current course of chemotherapy such that it dropped to <= 12 grams per deciliter) and baseline count of <125,000 microliters for developing red cells

Exclusion Criteria:

* Patients having a clinically significant disease other than cancer
* treated by platinum-containing chemotherapy within 3 months of study start
* having uncontrolled high blood pressure, a history of seizure, or untreated iron, folate, or Vitamin B12 deficiency
* received a transfusion or radiotherapy within 2 weeks of study start, or had surgery within 1 week of study start
* intending to use steroid drugs during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 1996-08; Study Completion 1998-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients transfused after one month

SECONDARY OUTCOMES:
Changes in hemoglobin, hematocrit, and developing red blood cells from the start of the study until study completion; Changes in quality-of-life; Safety

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Epoetin alfa for anemia in patients with cancer receiving non-platinum chemotherapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=684&filename=CR005917_CSR.pdf